CLINICAL TRIAL: NCT07321990
Title: Study of the Reproducibility of the French Version of the Modified SMAFRS Scale
Acronym: mSMAFRS-F
Status: Recruiting | Type: Observational
Sponsor: Institut de Myologie, France (Other)
Responsible Party: Sponsor
Other Study IDs: mSMAFRS-F
Record Dates: First submitted 2025-12-12; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: SMA
Keywords: SMA; Questionnaire; Translation; Validation
MeSH Terms: interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treated patients
  Interventions: Other: Questionnaire and Physical Exam

INTERVENTIONS:
Other: Questionnaire and Physical Exam — Patients will answer the french mSMA-FRS during their introduction to treatment or treatment follow-up visit, then again, fifteen days after this visit.
  Other Names: SMA-FRS

SUMMARY:
The goal of this observational study is to evaluate the test-retest reliability of the French version of the mSMAFRS in adult patients with SMA. The main question[s] is to answer if:

* ICC is a good estimate of test-retest reliability?
* mSMAFRS-F correlate with other outcome measures?

Participants will simply answer a french version of the SMA-FRS questionnaire during their routine follow-up visit then again fifteen days later.

DETAILED DESCRIPTION:
The modified SMAFRS is a patient-reported outcome measure (PROM) designed to assess the level of independence in ten activities of daily living (ADLs) within one's own environment for individuals with SMA. Activities include eating, dressing, bathing, toileting, grooming, turning in bed/adjusting bedclothes, transfers, walking, climbing stairs, and respiratory status. Each item is scored from 0 (fully dependent) to 5 (fully independent) by the patient or caregiver, maximum score of 40. The mSMAFRS has been used in several therapeutic and 9/21 2025-A00536-43_PROTOCOLE_V1.2_20250707_mSMAFRS-F observational studies. Feasibility, test-retest reliability, construct & content validity has been demonstrated for the English version. However currently no French version exists. Therefore, each clinician or health professional translates the items themselves during consultation with patients. This has consequences for inter-rater reliability as translations are likely to differ from one clinician to another and for intra-rater reliability as translations may differ at each visit. Therefore, successive evaluations are compromised. It is essential that an official French version exists for both clinical and research use. The added benefit of the mSMAFRS to other functional scales (e.g., MFM) is its specificity in SMA and its simplicity to perform as it is patient-reported and not observer-rated. It is useful and relevant for both ambulant and non-ambulant individuals and it includes a respiratory item which is lacking in the other functional scales.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Genetically confirmed SMA
* Able to comply with all protocol requirements (no significant cognitive impairment)
* French-speaking
* Affiliated or beneficiary of a social security scheme

Exclusion Criteria:

* Persons subject to a legal protection measure
* Subjects unable to complete the French version of the questionnaire mSMAFRS-Fbecause of lack of French fluency
* Subjects unable to complete the French version of the questionnaire mSMAFRS-Fbecause of cognitive impairment
* Inability to comply with protocol requirements
* Any medical and social conditions that could interfere with the study under theappreciation of the medical coordinator

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will be conducted in 60 adult's patients with SMA ≥18 years (ambulatory or not, treatment naïve or not).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Test-retest reliability | up to 2 weeks
  ICC is a good estimate of test-retest reliability. It is expected that mSMAFRS-F is highly reliable (ICC>0.9).

CONTACTS AND LOCATIONS:
Locations (1):
- Association institut de Myologie, Paris, France